CLINICAL TRIAL: NCT05773248
Title: Implementation of an Enhanced Recovery After Surgery (ERAS) Program in Colorectal Surgery: the Benefits of Late Adoption
Brief Title: ERAS in Colorectal Surgery: Benefits of Late Adoption
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-00221
Record Dates: First submitted 2023-02-13; First posted 2023-03-17 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Colorectal Cancer; Colorectal Neoplasms; Colorectal Disorders
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Standard care
- ERAS
  Interventions: Procedure: ERAS protocol

INTERVENTIONS:
Procedure: ERAS protocol — The main concepts of the ERAS protocol compared to standard care included the following aspects: preoperative counselling with a specially trained nurse, restrictive use of preoperative sedation, intraoperative fluid and opioid administration and drain placement, strict antiemetic prophylaxis, early mobilisation, bowel stimulation and removal of any catheters as well as early food intake. Additionally, the ERAS protocol included a 30-day telephone follow-up.
  Groups: ERAS

SUMMARY:
The aim of this single-center retrospective cohort study is to explore the effect of late adaptation of an ERAS protocol in a high-volume colorectal surgical unit.

The primary endpoint is the surgical outcome measured by early postoperative complications, defined by the comprehensive complications index. Secondary endpoints include amongst others LOS (length of stay), cost analysis, short-term follow-up in the ERAS group.

DETAILED DESCRIPTION:
At Clarunis - University Center for Gastrointestinal and Liver Diseases at St. Claraspital between 2019 und 2020, all colorectal patients were treated according to a standardized perioperative protocol. As of 2021 until today, an ERAS protocol was established and all colorectal patients who met inclusion criteria participated in this program automatically as part of a new standardized care. Perioperative data was collected in a clinical information system (Phoenix - CGM Clinica Information Systeml).

In this retrospective cohort study, we compare demographic, perioperative and postoperative data among the two groups "ERAS" and "non-ERAS" using a weighted propensity score analysis for patients who underwent surgery as part of the ERAS program and for patients without a standardized ERAS protocol.

All patients treated at the colorectal unit from 2019 until August 2022 and who are considered for the analysis have given written general consent for the use of health-related data for research projects (attached to this document).

ELIGIBILITY:
Inclusion Criteria:

* written general informed consent
* patients undergoing a colorectal procedure between 2019 and August 2022 at colorectal unit, Santa Clara Hospital, Basel

Exclusion Criteria:

* All patients undergoing an emergency procedure or a combined procedure with the colorectal procedure not being the main indication for surgical treatment (i.e. gynecological debulking, liver resection, etc.) were excluded from the analysis.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing a colorectal procedure between 2019 and August 2022 at colorectal unit, Santa Clara Hospital, Basel
Sampling Method: Non-Probability Sample
Enrollment: 456 (Actual)
Dates: Start 2023-03-13 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Perioperative morbidity | 30days
  Postoperative complications according to the comprehensive complication index (CCI)

SECONDARY OUTCOMES:
Length of stay | 30 days up to 3 months
  Length of postoperative hospital stay (days)
Cost analysis | 30 days up to 3 months
  All costs and incomes for every single case is assessed to calculate the loss or revenue. This data is obtained from the in-hospital financial department.
  If a patient is readmitted for a complication within 30 days, the costs and incomes for the readmission is added to the case of the initial operation.
Readmission rate | 30 days
  Rate of readmission within 30 days after the operation

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Steinemann, PD Dr., Study Director — University Hospital, Basel, Switzerland
Locations (1):
- St. Clara Hospital, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No
Currently, there is no plan to shared IPD.

REFERENCES:
- [Derived] Susstrunk J, Mijnssen R, von Strauss M, Muller BP, Wilhelm A, Steinemann DC. Enhanced recovery after surgery (ERAS) in colorectal surgery: implementation is still beneficial despite modern surgical and anesthetic care. Langenbecks Arch Surg. 2023 Dec 13;409(1):5. doi: 10.1007/s00423-023-03195-7. PMID 38091109